CLINICAL TRIAL: NCT00569686
Title: Lovaza Therapy of Peripheral Arterial Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subject meeting criteria
Sponsor: University of Virginia (Other)
Collaborators: Reliant Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13107
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Peripheral Artery Disease
Keywords: PAD; peripheral artery disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Omacor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): treatment with lovaza
  Interventions: Drug: lovaza
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lovaza — lovaza 4 gm po daily
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
Sixty patients with mild-to-moderate PAD (ABI 0.4-0.9) and hypertriglyceridemia (>200 mg/dl) already treated with statins will be imaged at baseline and randomized to Lovaza and placebo for 12 months. MR imaging will be repeated at the end of the 12-month period.

We hypothesize that treatment of hypertriglyceridemia in patients with PAD with Lovaza will reduce atherosclerotic plaque volume in the superficial femoral artery (SFA) by 2% over 1 year compared to placebo. Secondary aims will be to show improved plaque characteristics (thickened fibrous cap, reduced lipid-rich necrotic core, improved exercise calf muscle perfusion using first-pass contrast enhanced MRI and improved exercise treadmill performance with Lovaza compared to matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, any ethnicity, ages 55-75
* Mild to moderate PAD (ankle brachial index (ABI) of 0.4-0.9 in either or both limbs)
* Symptomatic intermittent claudication in either or both limbs
* Hyperlipidemia treated with HMG-CoA reductase inhibition with persistent hypertriglyceridemia (triglycerides>200).

Exclusion Criteria:

* Patients with critical limb ischemia
* Moderate to severe chronic kidney disease (requiring hemodialysis or glomerular filtration rate (GFR) < 45 ml/min)
* Contraindication to MRI (pacemakers, defibrillators, intraocular metal, certain intracerebral aneurysm clips, etc.)
* Claustrophobia
* Known allergy to gadolinium chelates
* Patients with iron storage disease

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
treatment of hypertriglyceridemia in patients with PAD with Lovaza will reduce or prevent progression of atherosclerotic plaque volume in the superficial femoral artery (SFA) by 2% over 1 year as compared to placebo. | one year

SECONDARY OUTCOMES:
show improved plaque characteristics, improved exercise calf muscle perfusion using first-pass contrast enhanced MRI and improved | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kramer, MD, Principal Investigator — University of Virginia Health System
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States